CLINICAL TRIAL: NCT02398760
Title: Relationship Between Clinical Tests and Clinical Outcomes After Motor Control Exercises Intervention for Non-specific Chronic Low Back Patients
Brief Title: Relationship Between Clinical Tests and Clinical Outcomes After Motor Control Exercises Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Crystian Bitencourt Soares de Oliveira, Msc Student, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UEPJMF-5402
Record Dates: First submitted 2015-03-19; First posted 2015-03-26 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Low Back Pain
Keywords: Low Back Pain; Clinical Instability; Motor Control Exercises; Clinical Tests
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Motor Control Exercises (Experimental): (Costa LOP et al. 2009; Hodges PW et al. 2009)
  Interventions: Other: Motor Control Exercises

INTERVENTIONS:
Other: Motor Control Exercises — Subjects performed 8 weeks of motor control exercises intervention, 2 weekly 1 hour per session, instructed by trained physiotherapists to apply this program following a protocol developed in programs previously reported (Costa et al. 2009; Hodges et al. 2009). The first stage aims to improve the activity of muscles that have poor control and reduce overactivity of superficial muscles, previously assessed, through drawing in maneuver with feedback real-time ultrasound and via palpation. The second stage of the treatment involved more functional exercises, first using static and then dynamic tasks.

SUMMARY:
Nowadays, the research priority in low back pain area have been find subgroup of patients with the same characteristics that might achieve better outcomes in a specific intervention. However, even though the studies in this area have increased, questions of this nature remaining without an adequate answer, or with limited evidence. Therefore, the investigators propose to examine the ability of clinical tests, developed to assess alterations related to clinical lumbar instability, to identify subgroups of patients with non specific chronic low back pain that may have better outcomes after a motor control exercises intervention.

DETAILED DESCRIPTION:
Changes relative to clinical instability are well established in individuals with non specific chronic low back pain. However, in this population, these changes vary widely, characterizing them as an heterogenous group. Motor Control Exercises (MCE) aims to improve the impaired coordination of deep and superficial muscles of the trunk, to reestablish the stability of the lumbar spine reducing the common alterations in this population, and are associated with reduction of pain and disability of patients with non specific chronic low back pain. To specific assessment of the changes found in this population, clinical tests are often used: in the assessment to identify motor control alterations; during intervention as parameter for treatment progress (e.g. to increase exercises difficulty); and after intervention, to ensure that there was normalization of the motor control. There are several clinical tests to assess changes relative to clinical instability, such as: Clinical Classification Scale (CCS) to assess abdominal muscles and the coordination between superficial and deep trunk muscles; Clinical Test of Thoracolumbar Dissociation (CTTD) to assess anterior/posterior tilt while maintain a constant position of thoracolumbar junction; and the Prone Instability Test (PIT) and Passive Lumbar Extension Test (PLET) used to detect structural lumbar instability.

Therefore, primary objectives of this study are: to investigate the ability of clinical tests in predict clinical outcomes, pain and disability, in motor control exercises program, and to investigate the association of two or more tests to predict clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 60 years.
* non specific chronic low back (pain for more than 3 months) with pain intensity of at least 3 points measured by pain numerical rating scale (0-10) and disability of at least 6 points in the 24-item Roland Morris Disability Questionnaire (0-24).
* classified as low or medium risk though StarT Back Screening Tool

Exclusion Criteria:

* cardiovascular and neurological pathologies
* serious pathology in the spine and pelvic.
* previous spinal surgery of at least 1 year before the trial period.
* check-list with the red flags was performed to exclusion
* classified as high risk through StarT Back Screening Tool, due these patients have high psychological components and needed of specialized psychological attendance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pain (Numerical Rating Scale (0-10) | After Intervention (2 months), 6 months
Disability (measured by 24-item Roland Morris Disability Questionnaire) | After Intervention (2 months), 6 months
  Disability will be measured by 24-item Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
Function (Patient Specific Functional Scale (0-10) | After Intervention (2 months)
Global Perceived Effect (11-point Global Perceived Effect Scale (-5-+5) | After Intervention (2 months)
  11-point Global Perceived Effect Scale (-5-+5)
Depression (Beck Inventory (0-63) | After Intervention (2 months)
  Beck Inventory (0-63)
Kinesiophobia (Tampa Scale for Kinesiophobia (17-68) | After Intervention (2 months)
  Tampa Scale for Kinesiophobia (17-68)
Kinesiophobia (Fear Avoidance Beliefs Questionnaire (0-66) | After Intervention (2 months)
  Fear Avoidance Beliefs Questionnaire (0-66)
Kinesiophobia (Photograph Series of Daily Activities - Short Electronic Version (PHODA-SEV) (0-100) | After Intervention (2 months)
  Photograph Series of Daily Activities - Short Electronic Version (PHODA-SEV) (0-100)

OTHER OUTCOMES:
Clinical Classification Scale (CCS) | After Intervention (2 months)
  To assess abdominal muscles coordination (0-10)
Thoracolumbar Dissociation Clinical Test (TDCT) | After Intervention (2 months)
  To assess thoracolumbar dissociation (0-10)
Changes Thickness of abdominal muscles (Transversus Abdominis, Internal and External Oblique) Measured by Ultrasound Images | After Intervention (2 months)
  Measured by Ultrasound Images made with a 7.5-MHz linear transducer (Siemens, Sonoline Sienna, Issaquah, WA, USA)
Structural Lumbar Instability (Prone Instability Test (PIT) and Passive Lumbar Extension Test (PLET) | After Intervention (2 months)
  Prone Instability Test (PIT) and Passive Lumbar Extension Test (PLET)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben FN Filho, PhD, Principal Investigator — UNIVERSIDADE ESTADUAL PAULISTA JULIO DE MESQUITA FILHO
Locations (1):
- Centro de Atendimento em Reabilitação e Fisioterapia - FCT/UNESP, Presidente Prudente, São Paulo, Brazil

REFERENCES:
- [Background] Hodges PW, Ferreira PH, Ferreira ML. Lumbar spine: Treatment of instability and disorders of movement control. Magee DJ, Zachazewski JE, Quillen WS, editors. Pathology and Intervention in Musculoskeletal Rehabilitation. St. Louis: Saunders Elsevier. 2009;401
- [Background] Elgueta-Cancino E, Schabrun S, Danneels L, Hodges P. A clinical test of lumbopelvic control: development and reliability of a clinical test of dissociation of lumbopelvic and thoracolumbar motion. Man Ther. 2014 Oct;19(5):418-24. doi: 10.1016/j.math.2014.03.009. Epub 2014 Mar 30. PMID 24853256
- [Background] Hicks GE, Fritz JM, Delitto A, McGill SM. Preliminary development of a clinical prediction rule for determining which patients with low back pain will respond to a stabilization exercise program. Arch Phys Med Rehabil. 2005 Sep;86(9):1753-62. doi: 10.1016/j.apmr.2005.03.033. PMID 16181938
- [Background] Kasai Y, Morishita K, Kawakita E, Kondo T, Uchida A. A new evaluation method for lumbar spinal instability: passive lumbar extension test. Phys Ther. 2006 Dec;86(12):1661-7. doi: 10.2522/ptj.20050281. Epub 2006 Oct 10. PMID 17033040
- [Background] Bystrom MG, Rasmussen-Barr E, Grooten WJ. Motor control exercises reduces pain and disability in chronic and recurrent low back pain: a meta-analysis. Spine (Phila Pa 1976). 2013 Mar 15;38(6):E350-8. doi: 10.1097/BRS.0b013e31828435fb. PMID 23492976
- [Derived] Oliveira CB, Pinto RZ, Schabrun SM, Franco MR, Morelhao PK, Silva FG, Damato TM, Negrao Filho RF. Association Between Clinical Tests Related to Motor Control Dysfunction and Changes in Pain and Disability After Lumbar Stabilization Exercises in Individuals With Chronic Low Back Pain. Arch Phys Med Rehabil. 2019 Jul;100(7):1226-1233. doi: 10.1016/j.apmr.2019.01.019. Epub 2019 Feb 26. PMID 30822389